CLINICAL TRIAL: NCT02326129
Title: A Novel Biomarker for Development of Type 2 Diabetes: 11Beta-Hydroxy Steroid Dehydrogenase Type 1 Activity
Brief Title: Novel Biomarker for Development of T2D
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Children's Miracle Network (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00057460; K23DK117067 (NIH)
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 24 hour urine samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obese with Type 2 Diabetes: Obese adolescents with Type 2 Diabetes
- Obese without Type 2 Diabetes: Obese adolescents without Type 2 Diabetes
- Normal weight: Normal weight adolescents

SUMMARY:
The investigators wants to determine if 11β-HSD1 activity will be positively associated, and 5α-reductase activity negatively associated, with (a) degree of insulin resistance defined by the homeostatic model assessment of insulin resistance index (HOMA-IR) and (b) worsening glycemic control defined by higher HbA1c and impaired fasting glucose in a group of obese children and young adults with or without type 2 diabetes compared to lean children and young adults without diabetes. The investigators also want to identify key metabolic signatures associated with diabetes using metabolomic profiling.

DETAILED DESCRIPTION:
The overarching hypothesis is that increases in whole body 11β-HSD1 activity precede and presage the development of type 2 diabetes (T2D) in high-risk obese adolescents, serving as a critical determinant of insulin resistance and glucose intolerance. The increase in 11β-HSD1 activity, in combination with decreases in 5α-reductase activity, will increase tissue cortisol production, promoting the development of insulin resistance and the metabolic syndrome and predisposing to T2D. The investigators predict that increases in 11β-HSD1 activity will be detected in obese children prior to the development of insulin resistance and glucose intolerance and that the progressive increases in 11β-HSD1 will correlate with progressive decreases in insulin sensitivity and glucose tolerance. Given preliminary findings, the investigators also predict that increases in 11β-HSD1 will be greater and occur earlier in development in males than females. This could establish 11β-HSD1 activity as a novel, non-invasive biomarker for progression to, or for development of, glucose intolerance and T2D.

The identification of 11β-HSD1 as a biomarker that predicts T2D would have critical clinical import, allowing us to identify obese children and adults at highest risk of metabolic decompensation. Studies of 11β-HSD1 in obese subjects with varying degrees of IR and glucose intolerance will also narrow critical gaps in the understanding of the pathogenesis of T2D.

The investigators would like to also validate if urine metabolomic profiling can be used for identifying key metabolomic signatures associated with insulin resistance. To that end the investigators would like to examine detailed metabolomic profiles in 24 hour and spot urine samples.

The study population will include 50 obese adolescents with T2D, 50 obese adolescents without T2D and 50 age, gender, race and pubertal status-matched normal weight controls. The subjects will be recruited at the Healthy Lifestyle Program at Duke, Diabetes Clinics at Lenox Baker Children's Hospital and Roxboro Clinics.

Study activities include physical exam and medical history, vitals, laboratory tests (only for obese adolescents), urine testing for sugar (only for normal weight adolescents), 24 hour urine collection, spot urine collection, body fat content measurement, and food and activity questionnaire.

ELIGIBILITY:
Inclusion criteria:

1. Obese/Overweight adolescents/young adults without T2D who are having their first visit to the Healthy Lifestyle Program at Duke or Obese/Overweight adolescents/young adults without T2D recruited from the community at PBRC
2. Obese/Overweight adolescents/young adults with prediabetes (HbA1c between 5.7-6.4%) and T2D (HbA1c≥6.5%)followed at Diabetes Clinics or recruited from the community at PBRC
3. Age, gender, race and pubertal status matched normal weight adolescents presenting for "well child check" at Roxboro Clinics
4. ≥12 to 21 (inclusive) years of age for urine studies
5. 18-21 years of age obese adolescents/young adults without T2D and age, gender, race and pubertal status matched normal weight controls for OGTT sub-study
6. Both the subject and one parent/guardian present will need to be able to speak and read English

Exclusion criteria:

1. Currently or within the past month taken systemic or inhaled corticosteroids, antipsychotics, medications for weight loss, topiramate, acute use of contraceptives (less than 3 months) or medroxy-progesterone acetate, medications to treat ADHD
2. Children with any genetic syndrome
3. Children with decompensated hypothyroidism (treated with levothyroxine and a TSH >10 µIU/mL )
4. Normal weight children (BMI percentile 5%-<85%) with glucosuria, as defined by a positive urine glucose dip stick test
5. Children and young adults who self report that they are pregnant (pregnancy is excluded in both the main and sub-study)
6. Proteinuria, as defined by protein level equal to or above 300 mg/dl (+++) on a urine dip stick test.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will include 50 obese adolescents with Type II Diabetes, 50 obese adolescents without Type II Diabetes, and age, gender, race and pubertal status-matched normal weight controls for urine study and 32 young adults 18-21 years of age obese adolescents without T2D and age, gender, race and pubertal status matched normal weight controls for OGTT sub-study.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2015-02; Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Relationship between 11β-HSD1 and 5α-reductase activity, and measures of insulin resistance | One year
  To assess the relationship between 11β-HSD1 and 5α-reductase activity, and measures of insulin resistance in a cohort of obese children with varying degrees of insulin resistance and glucose intolerance
Gender and pubertal status | One year
  Investigate the role of gender and pubertal status on 11β-HSD1 and 5α-reductase activity
Compare 11β-HSD1 activity and 5α-reductase activity among obese adolescents with T2D, obese adolescents without T2D and normal weight controls | One year
  The investigators hypothesize that obese adolescents with T2D will have the highest levels of 11β-HSD1 activity followed by the obese adolescents with insulin resistance, followed by obese subjects with normal insulin sensitivity. Normal weight control group will have the lowest levels.

SECONDARY OUTCOMES:
Relationship between 11β-HSD1 and 5α-reductase activity, and key metabolic signatures associated with insulin resistance | One year
  The investigators hypothesize that 11β-HSD1 activity will be positively associated, and 5α-reductase activity negatively associated, with key metabolic signatures associated with insulin resistance.
Urine metabolic signatures associated with insulin resistance and type 2 diabetes | One year
  The investigators would like to validate if urine metabolomic profiling can be used for identifying key metabolomic signatures associated with insulin resistance
Spot urine for metabolic profiling | One year
  The investigators hypothesize that they will identify the same key metabolomic signatures associated with insulin resistance in obese adolescents with T2D compared to obese adolescents without T2D, and normal weight control group in spot fasting am urine samples.
Metabolic signatures correlate with parameters of glucose tolerance | One year
  To determine if urinary metabolic signatures correlate with parameters of glucose tolerance in normal weight controls and obese adolescents without T2D, and glycemic control in obese subjects with T2D.

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Gumus Balikcioglu, M.D., Principal Investigator — Pediatric Endocrinology
Locations (3):
- United States (3):
  - Pennington Biomedical Research center, Baton Rouge, Louisiana
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina